CLINICAL TRIAL: NCT03003364
Title: A Phase I/IIa, Randomized, Double-blind, Single-dose, Placebo Controlled, Two-way Crossover Clinical Trial to Assess the Safety and to Obtain Efficacy Data in Intrathecal Administration of Expanded Wharton's Jelly Mesenchymal Stem Cells in Chronic Traumatic Spinal Cord Injury
Brief Title: Intrathecal Administration of Expanded Wharton's Jelly Mesenchymal Stem Cells in Chronic Traumatic Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Hospital de Neurorehabilitació Institut Guttmann (Unknown); Recerca Clínica S.L. (Industry); Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XCEL-SCI-01
Record Dates: First submitted 2016-12-14; First posted 2016-12-28 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injury, Chronic
MeSH Terms: conditions — Spinal Cord Injuries; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XCEL-UMC-BETA/placebo (Experimental): Ex vivo cultured human mesenchymal stem cells from Wharton jelly, in a blinded syringe (initial treatment) / Placebo (month 6)
  Interventions: Drug: XCEL-UMC-BETA; Drug: Placebo
- Placebo/XCEL-UMC-BETA (Placebo Comparator): Placebo in a blinded syringe (initial treatment) / XCEL-UMC-BETA (month 6)
  Interventions: Drug: XCEL-UMC-BETA; Drug: Placebo

INTERVENTIONS:
Drug: XCEL-UMC-BETA — Intrathecal allogeneic cell therapy in a blinded syringe
  Other Names: Expanded MSC from Wharton Jelly
Drug: Placebo — Placebo in a blinded syringe

SUMMARY:
This is a phase I/IIa, randomized, double-blind, two-arms, two-dose administration, placebo controlled, two-way crossover clinical trial in which 10 patients from 18 to 65 years of age affected with chronic traumatic spinal cord will enter the study with the objective to assess the safety and to obtain efficacy data in intrathecal administration of expanded Wharton's jelly mesenchymal stem cells.

DETAILED DESCRIPTION:
This is a phase I/IIa, randomized, double-blind, two-arms, two-dose administration, placebo controlled, clinical trial in which 10 patients from 18 to 65 years of age affected with chronic traumatic spinal cord will enter the study with the objective to assess the safety and to obtain efficacy data in intrathecal administration (L3 level) of expanded Wharton's jelly mesenchymal stem cells. Following the administration patients will remain for 24 h at the hospital and thereafter will be discharged. For the first period, the follow-up is planned at day 7 and at 1, 3 and 6 months. At month 6, the patients will be treated in a crossover way (second period) and will follow the same schedule for the follow-up. First clinical trial evaluation will be performed at 12 month follow-up. From 12 to 18 month after the first infusion, patients will be randomized again to active treatment or placebo (double-blind) in order to assess the safety and efficacy of a second dose at 12 month follow-up. Thereafter, patients will be followed up at 24 and 36 months as part of a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Single spinal cord injury lesion caused by trauma
2. Affected cord segments between T2 and T11, confirmed by magnetic resonance
3. Complete paraplegia (ASIA A)
4. Chronic disease state (between 12 months and 5 years after the injury)
5. Patients from 18 to 65 years of age, both sexes
6. Life expectancy > 2 years
7. Confidence that the patient will attend the follow-up visits.
8. Given informed consent in writing
9. Patient is able to understand the study and its procedures

Exclusion Criteria:

1. Mechanic ventilation
2. Lesion affecting multiple levels
3. Lesion length superior to 3 spinal cord segments, assessed by magnetic resonance
4. Penetrating trauma affecting the spinal cord
5. Positive serology to HIV, HBV, HCV and or syphilis
6. Pregnant woman or without proper anticonceptive measures according to the investigator, or breath feeding
7. Use of metal implants that complicates the MRI interpretation
8. Planned spinal surgery within subsequent 24 month after entering the trial
9. Intrathecal medication or immunosuppressive drugs the previous 60 days.
10. Neurodegenerative diseases
11. Significant abnormal laboratory tests that contraindicates patient's participation in the study.
12. Neoplasia within the previous 5 years, or without complete remission
13. Patient with difficulty for communicating
14. Participation in another clinical trial or treated with an investigational medicinal product the previous 60 days
15. Contraindication for lumbar punction
16. Other pathologic conditions or circumstances that could complicate the participation of the patient in the study according to medical criteria
17. The patient does not accept to be followed-up for a period that could exceed the clinical trial length

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 12 months
  Adverse events

SECONDARY OUTCOMES:
Extent and severity of a patient's spinal cord injury | 6 months
  ASIA Impairment Scale
Motor electrophysiology assessment | 6 month
  Evoked potentials
Somatosensory electrophysiology assessment | 6 month
  Evoked potentials
Electrical nerve stimulation on pain perception | 6 month
  Pain threshold perception
Mictional dysfunction | 6 month
  Urodynamic testing
Anal sphincter integrity | 6 month
  Anorectal manometry test
Neuropathic pain | 6 months
  Numerical scale (0 to 10)
Spasticity | 6 months
  Modified Ashworth scale
Functionality | 6 months
  SCIM III scale
Quality of life (individual overall perception of quality of life, individual overall perception of their health, Physical health, Psychological, Social relationships, Environment) | 6 months
  WHOQOL BREF questionnaire
Urinary disorder | 6 months
  Qualiveen questionnaire
Size injury | 12 months
  Magnetic Resonance Imaging
Presence of allogeneic cells | 1 month
  Chimerism in cerebrospinal fluid
Immunology | 1 months
  Antibodies anti-HLA in peripherical blood and in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Joan Vidal, MD, PhD, Principal Investigator — Hospital de Neurorehabilitació Institut Guttmann
Locations (1):
- Hospital de Neurorehabilitació Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albu S, Kumru H, Coll R, Vives J, Valles M, Benito-Penalva J, Rodriguez L, Codinach M, Hernandez J, Navarro X, Vidal J. Clinical effects of intrathecal administration of expanded Wharton jelly mesenchymal stromal cells in patients with chronic complete spinal cord injury: a randomized controlled study. Cytotherapy. 2021 Feb;23(2):146-156. doi: 10.1016/j.jcyt.2020.08.008. Epub 2020 Sep 25. PMID 32981857
- See also: Hospital de Neurorehabilitació Institut Guttmann — http://www.guttmann.com/en
- See also: Marató TV3 — http://www.ccma.cat/tv3/marato/en/